CLINICAL TRIAL: NCT02452749
Title: Prospective Safety and Tolerability Assessment of a Cardiovascular Health Dietary Supplement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Natural Medicine (Other)
Responsible Party: Principal Investigator, Jennifer Ryan, Postdoctoral Fellow, National University of Natural Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRB042115
Record Dates: First submitted 2015-05-19; First posted 2015-05-25 (Estimated); Last update posted 2018-03-15 (Actual); Status verified 2018-03

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cardiovascular Health Dietary Supplement (Experimental): The cardiovascular health dietary supplement will be administered at a dosage of 1 caplet po per day for a period of 6 months
  Interventions: Dietary Supplement: Cardiovascular health dietary supplement

INTERVENTIONS:
Dietary Supplement: Cardiovascular health dietary supplement — Herbal/mineral dietary supplement

SUMMARY:
This single-arm, open-label study will assess the safety and tolerability of one daily tablet of a commercially available cardiovascular health dietary supplement by questionnaire and blood markers in adults with borderline to mild hypertension over a 6 month period. Although the cardiovascular health dietary supplement being investigated has been on the market for over 20 years, prospective safety data and blood markers of end organ function have not previously been reported.

DETAILED DESCRIPTION:
Hypertension is an important overall risk factor for developing cardiovascular disease in the United States, and is a leading risk factor for cardiovascular events, including myocardial infarction and stroke, and cardiovascular-related mortality with advancing age. Based on population based studies and clinical trials, both systolic blood pressure (SBP) and diastolic blood pressure (DBP) elevations are continuous, strong and independent risk factors for cardiovascular disease.

The product being studies is a cardiovascular health dietary supplement that has been commercially available since 1993. It is currently sold to healthcare practitioners as well as directly to consumers. Some healthcare providers use the product as part of a plan to treat high blood pressure in their patients. This is the first study collecting prospective safety data on this product.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65
* Systolic blood pressure 120-159 mmHg or diastolic blood pressure 80-99 mmHg upon screening

Exclusion Criteria:

* Bradycardia
* Initiation of or changes to blood pressure lowering medications within the last month
* Initiation of or changes to thyroid medications within the last month
* Currently taking any of the following orally (or they were taken within the last month):

  * Rauwolfia serpentina, Terminalia arjuna, Tribulus terrestris, Convolvulus pluricaulis, Boerhavia diffusa, Rosa vinca, rose powder, or coral powder
  * Beta blockers
  * Alpha blockers
  * Propranolol
  * Digoxin
  * Levodopa
  * Anti-depressant medications
  * Anti-psychotic medications
  * Sedatives or tranquilizers
* Present or past history of any of the following:

  * Cardiovascular disease
  * Heart surgery
  * Cardiac arrhythmia
  * Abnormal EKG
  * Abnormal echocardiogram
  * Diabetes
  * Chronic liver, kidney or bowel disease
  * Ulcers
  * Gallbladder disease
  * Depression
  * Alcoholism
  * Obstructive sleep apnea and/or use of a continuous positive airway pressure device
  * Parkinson's disease
  * Pheochromocytoma
  * Cancer within the last 5 years
* Consuming more than fourteen alcoholic beverages per week
* Current smoking/tobacco use
* Current illicit and/or recreational drug use
* Women who are lactating, pregnant or planning pregnancy within the next six months
* Known intolerance or allergy to study agents

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-05-01 (Actual); Primary Completion 2017-07-28 (Actual); Study Completion 2017-07-28 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of a cardiovascular health dietary supplement assessed by composite changes in multi-system symptoms, a validated mood/depression questionnaire, electrolytes, and surrogate markers of heart, liver and kidney function | Baseline, 3 months, 6 months
  Standardized adverse event monitoring form, Patient Health Questionnaire (PHQ-9), electrolytes (sodium, potassium, calcium, magnesium), b-type natriuretic peptide, aspartate aminotransferase, alanine aminotransferase, and estimated glomerular filtration rate

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer J Ryan, ND, MS, Principal Investigator — National University of Natural Medicine
Locations (1):
- Helfgott Research Institute, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No